CLINICAL TRIAL: NCT02688946
Title: Imaging Microcirculation And Gross Hemodynamic Assessment of the Bowel During Elective Colorectal Surgery
Brief Title: Imaging Microcirculation and Gross Hemodynamics in Elective Colorectal Surgery
Acronym: IMAGES
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, Coordinating investigator, St. Antonius Hospital
Other Study IDs: NL4833210014
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Microcirculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not provided

SUMMARY:
Rationale: The interaction between macro and microcirculation remains uncertain. Microvascular alterations can occur when systemic hemodynamic parameters are within an acceptable range. Perfusion changes and microvascular alterations may play an important role in anastomotic healing and the onset of anastomotic leakage after gastrointestinal surgery. Nowadays, assessment of bowel perfusion is macroscopically performed by the surgeon prior to anastomosis creation. However, local oxygen delivery may still be compromised as little is known about microcirculatory alterations of the bowel during colorectal surgery. Dark Field (DF) imaging is a technique using a stroboscopic light-emitting diode ring-based imaging modality incorporated in a hand-held device, which illuminates an area of interest and provides high contrast dynamic images of the microvasculature. DF-imaging enables to visualize the bowel's microcirculation.

Objective: To describe the human gastrointestinal microcirculation during gastrointestinal surgery under general anesthesia and to observe whether there is a correlation between bowel microcirculation and systemic hemodynamic parameters.

Study design: A prospective, single center, observational, clinical, pilot study.

Study population: 70 patients undergoing elective, gastrointestinal surgery during which the gastrointestinal tract is accessible for DF-imaging.

Main study parameters/endpoints: To describe human gastrointestinal microcirculation on both the serosal and mucosal side of the bowel during gastrointestinal surgery under general anesthesia. Main parameter: Microvascular perfusion is quantified using the Microvascular Flow Index (MFI).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The extend of burden and risk associated with participation is negligible. Using DF imaging on the bowel is a non-invasive technique requiring a minimal amount of time as is described in the study procedure. Previous studies did not show any safety concerns. Measuring will be performed under sterile conditions and the occurrence of tissue damage is highly unlikely. Patients are under general anesthesia and will thus not experience any inconvenience.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 scheduled for elective, gastrointestinal surgery (as described above) with signed informed consent.

Exclusion Criteria:

* • Age <18 years;

  * Atrial fibrillation (because of possible interference with FloTrac™/Vigileo™ cardiac output monitor);
  * Left ventricular ejection fraction ≤30%;
  * Serious pulmonary disease (resting pO2 <90% at room air);
  * Renal failure (clearance <30 ml/min as calculated using the Modification of Diet in Renal Disease formula);
  * Liver failure;
  * No signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients undergoing elective, gastrointestinal surgery. Surgical procedures included will be:
  * All forms of open colorectal surgery;
  * Pylorus Persevering PancreaticoDuodenectomy (PPPD);
  * Other procedures requiring small bowel resection for cancer;
  * Laparoscopic procedures with extracorporeal creation of the bowel anastomosis. These procedures provide unique access to different parts of the bowel. The PPPD procedure provides access to the mucosal and serosal side of the jejunum. Colorectal surgery provides access to both the serosal and mucosal side of the colon and the terminal ileum is sometimes also accessible. We expect to include around 2 patients per week.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index (MFI) | Intra-operative
  During surgery

SECONDARY OUTCOMES:
Perfused vessel density (PVD) | Intra-operative
Proportion of perfused vessels (PPV) | Intra-operative
Total vessel density (TVD) | Intra-operative
Heterogeneity index (HI) | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mat Van Iterson, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tavy ALM, de Bruin AFJ, van der Sloot K, Boerma EC, Ince C, Noordzij PG, Boerma D, van Iterson M. Effects of Thoracic Epidural Anaesthesia on the Serosal Microcirculation of the Human Small Intestine. World J Surg. 2018 Dec;42(12):3911-3917. doi: 10.1007/s00268-018-4746-z. PMID 30097706